CLINICAL TRIAL: NCT02953743
Title: Pharmacokinetic Study of E7080/Lenvatinib in Chinese Patients With Unresectable Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-C086-107
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-02

CONDITIONS: Unresectable Hepatocellular Carcinoma (HCC)
Keywords: E7080; Lenvatinib; Pharmacokinetic study; Chinese participants; Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lenvatinib 12 mg (Experimental): Participants weighing ≥ 60 kg will be enrolled in this arm.
  Interventions: Drug: Lenvatinib
- Lenvatinib 8 mg (Experimental): Participants weighing < 60 kg will be enrolled in this arm.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — Lenvatinib 4 mg capsules will be administered orally, once daily continuously 28-day cycles until disease progression, development of unacceptable toxicity or withdrawal of consent.

SUMMARY:
The primary purpose of this study is to assess the single- and multiple-dose pharmacokinetic (PK) profile of lenvatinib in Chinese participants with unresectable Hepatocellular Carcinoma (HCC).

ELIGIBILITY:
Inclusion Criteria

1. Participants must have confirmed diagnosis of unresectable Hepatocellular Carcinoma (HCC) with any of the following criteria:

   1. Histologically or cytologically confirmed diagnosis of HCC
   2. Clinically confirmed diagnosis of HCC according to American Association for the Study of Liver Diseases (AASLD) criteria, including cirrhosis of any etiology or with chronic hepatitis B or C infection criteria
2. Participants categorized to stage B (not applicable for transarterial chemoembolization [TACE]) or stage C based on Barcelona Clinic Liver Cancer (BCLC) staging system
3. Adequate bone marrow function, defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/Liter (L)
   2. Hemoglobin (Hb) ≥ 8.5 gram per deciliter (g/dL)
   3. Platelet count ≥ 75 × 10^9/L
4. Adequate liver function, defined as:

   1. Albumin ≥ 2.8 g/dL
   2. Bilirubin ≤ 3.0 milligram per deciliter (mg/dL)
   3. Aspartate aminotransferase (AST), alkaline phosphatase (ALP), and alanine aminotransferase (ALT) ≤ 5 × the upper limit of normal (ULN)
5. Adequate blood coagulation function, defined as international normalized ratio (INR) ≤ 2.3
6. Adequate renal function defined as creatinine clearance > 40 milliliter per min (mL/min) calculated per the Cockcroft-Gault formula
7. Adequately controlled blood pressure (BP) with up to 3 antihypertensive agents, defined as systolic BP ≤ 150 millimeter of mercury (mm Hg) and diastolic BP ≤ 90 mm Hg at screening and no change in antihypertensive therapy within 1 week prior to the registration.
8. Child-Pugh A (score 5-6)
9. Eastern Cooperative Oncology Group (ECOG)- performance status (PS) 0 or 1
10. Survival expectation of 12 weeks or longer after starting study drug
11. Males or females aged at least 18 years at the time of informed consent.
12. Females must not be lactating or pregnant at Screening or Baseline (as documented by a negative beta-human chorionic gonadotropin [Beta-hCG] test with a minimum sensitivity of 25 International Unit/Liter [IU/L] or equivalent units of beta-hCG). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.
13. All females will be considered to be of childbearing potential unless they are postmenopausal (amenorrheic for at least 12 consecutive months, in the appropriate age group and without other known or suspected cause) or have been sterilized surgically (ie, bilateral tubal ligation, total hysterectomy or bilateral oophorectomy, all with surgery at least one month before dosing).
14. Females of childbearing potential must not have had unprotected sexual intercourse within 30 days before study entry and must agree to use a highly effective method of contraception (eg, total abstinence, an intrauterine device, a double-barrier method [such as condom plus diaphragm with spermicide], a contraceptive implant, an oral contraceptive, or have a vasectomized partner with confirmed azoospermia) throughout the entire study period and for 30 days after study drug discontinuation. If currently abstinent, the participant must agree to use a double barrier method as described above if she becomes sexually active during the study period or for 30 days after study drug discontinuation. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks before dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
15. Male participants must have had a successful vasectomy (confirmed azoospermia) or they and their female partners must meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period and for 30 days after study drug discontinuation). No sperm donation is allowed during the study period and for 30 days after study drug discontinuation.
16. Provide written informed consent
17. Willing and able to comply with all aspects of the protocol as judged by the Investigator.

Exclusion Criteria

1. Imaging findings for HCC corresponding to any of the following:

   1. HCC with ≥50% liver occupation
   2. Clear invasion into the bile duct
   3. Portal vein invasion at the main portal branch (Vp4)
2. Participants who have received lenvatinib
3. Participants who have received any anti-cancer therapy (including surgery, percutaneous ethanol injection, radio frequency ablation, transarterial [chemo] embolization, hepatic intra-arterial chemotherapy, biological, immunotherapy, hormonal, any investigational drugs or radiotherapy) or any blood enhancing treatment (including blood transfusion, blood products, or agents that stimulate blood cell production, eg, granulocyte colony-stimulating factor [G-CSF]) within 28 days prior to registration.
4. Participants who have not recovered from toxicities as a result of prior anticancer therapy except alopecia and infertility. Recovery is defined as < Grade 2 severity per Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4.0).
5. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at screening
6. Prolongation of Q wave and T wave interval corrected by the Fridericia formula (QTcF) interval to > 480 milli second (msec)
7. Gastrointestinal malabsorption, or any other condition in the opinion of the investigator that might affect the absorption of lenvatinib
8. Bleeding or thrombotic disorders or use of anticoagulants requiring therapeutic INR monitoring, eg, warfarin or similar agents. Treatment with low molecular weight heparin and factor X inhibitors which do not require INR monitoring is permitted. Antiplatelet agents are prohibited throughout the study.
9. Gastrointestinal bleeding event within 28 days prior to registration
10. Gastric or esophageal varices that require interventional treatment within 28 days prior to randomization. Prophylaxis with pharmacologic therapy (eg, nonselective beta-blocker) is permitted.
11. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 28 days prior to registration
12. Active malignancy (except for HCC or definitively treated melanoma in-situ, basal or squamous cell carcinoma of the skin, or carcinoma in-situ of the cervix) within the past 36 months from registration.
13. Any history of or current brain or subdural metastases
14. Participants having > 1+ proteinuria on urine dipstick testing will undergo 24h urine collection for quantitative assessment of proteinuria. Participants with urine protein ≥ 1 gram (g)/24 hour (h) will be ineligible.
15. Surgical arterial-portal venous shunt or arterial-venous shunt.
16. Any medical or other condition that in the opinion of the investigator would preclude participation in a clinical study
17. Human immunodeficiency virus (HIV) positive, or active infection requiring treatment (except for hepatitis virus)
18. History of drug or alcohol dependency or abuse within approximately 2 years prior to registration.
19. Any participant who cannot be evaluated by dynamic CT because of allergic reaction to contrast agent of CT.
20. Major surgery within 3 weeks prior to registration or scheduled for surgery during the study
21. Participant who has had a liver transplant.
22. Participants whose only tumor lesion(s) is in bone will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-06-28 (Actual); Study Completion 2020-12-28 (Actual)

PRIMARY OUTCOMES:
Mean maximum observed concentration (Cmax) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose
Mean time at which the highest drug concentration occurs (tmax) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose
Mean area under the concentration-time curve from zero time to time of last quantifiable concentration (AUC(0-t)) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose
Mean maximum observed concentration at steady-state (Css,max ) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose
Mean minimum observed concentration at steady-state (Css,min) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose
Average steady-state concentration (Css,av) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose
Mean time at which the highest drug concentration occurs at steady-state (tss,max) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose
Mean area under the concentration-time curve over the dosing interval on multiple dosing (AUC(0-τ)) | Day 1 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 2 at pre-dose; Day 8 at pre-dose; Day 15 at pre-dose, 0.5, 1, 2, 4, 6, and 8 hours; Day 16 at pre-dose; and Day 22 at pre-dose

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) and serious adverse events (SAEs) | Up to 30 days after the administration of the last dose of study drug or up to approximately 1 year

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Shanghai Cancer Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Bai Y, Hu X, Ren Z, Hisai T, Yusa W, Weng L, Shiba S, Takase T. A phase I pharmacokinetic study of lenvatinib in Chinese patients with unresectable hepatocellular carcinoma. Future Oncol. 2022 Jul;18(22):2413-2424. doi: 10.2217/fon-2022-0229. Epub 2022 Jun 8. PMID 35674480